CLINICAL TRIAL: NCT00387933
Title: Phase I Dose Escalation of Gleevec in Combination With PTK787/ZK 222584 (PTK/ZK) Plus Hydroxyurea
Brief Title: Imatinib Mesylate, Vatalanib, and Hydroxyurea in Treating Patients With Recurrent or Relapsed Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00006014; DUMC-7019-06-3R1; NOVARTIS-DUMC-7019-06-3R1
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2012-11

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult gliosarcoma; adult giant cell glioblastoma; adult anaplastic ependymoma; adult brain stem glioma; adult mixed glioma; adult pineal gland astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Gliosarcoma; Ependymoma; Glioma | interventions — Hydroxyurea; Imatinib Mesylate; vatalanib

ARMS (1):
- Gleevec + PTK787/ZK 22584 + Hydroxyurea (Experimental): Patients with recurrent or relapsing glioblastoma multiforme (GBM) will be given daily doses of Gleevec and PTK787/ZK 22584 orally in combination with fixed doses of hydroxyurea.
  Interventions: Drug: hydroxyurea; Drug: imatinib mesylate; Drug: vatalanib

INTERVENTIONS:
Drug: hydroxyurea
  Other Names: HU; hydrea
Drug: imatinib mesylate
  Other Names: Gleevec
Drug: vatalanib
  Other Names: PTK787

SUMMARY:
RATIONALE: Imatinib mesylate, vatalanib, and hydroxyurea may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Vatalanib may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving imatinib mesylate and vatalanib together with hydroxyurea may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of imatinib mesylate and vatalanib when given together with hydroxyurea in treating patients with recurrent or relapsed malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and dose-limiting toxicity of imatinib mesylate and vatalanib when administered with hydroxyurea in patients with recurrent or relapsed grade 3 or 4 malignant glioma.
* Determine the safety and tolerability of this regimen in these patients.
* Determine the single-dose and repeated-dose pharmacokinetic profiles of imatinib mesylate (in serum) and vatalanib in these patients.
* Determine the pre- and post-treatment antiangiogenic effects of this regimen in these patients, using dynamic contrast-enhanced MRI to evaluate changes in the extent of vascular permeability, perfusion, and relative tumor blood volume.
* Determine whether changes in diffusion-weighted images MRI (quantitated by apparent diffusion coefficient maps) correlate with tumor cellularity and tumor cell death in patients treated with this regimen.
* Determine antitumor activity of this regimen, in terms of radiographic response, progression-free survival, and overall survival, in these patients.

OUTLINE: This is an open-label, dose-escalation study of imatinib mesylate and vatalanib.

Patients receive oral vatalanib once daily, oral imatinib mesylate once daily, and oral hydroxyurea twice daily on days 1-28*. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients receive vatalanib alone daily on days 1-7 followed by vatalanib, imatinib mesylate, and hydroxyurea on days 8-35 in course 1 only.

Cohorts of 3-6 patients receive escalating doses of imatinib mesylate and vatalanib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

After completion of study treatment, patients will be evaluated for 28 days.

PROJECTED ACCRUAL: A total of 42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant glioma

  * Grade 3 or 4 disease
  * In first, second, or third recurrence or relapse
* Multifocal disease allowed

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Life expectancy ≥ 12 weeks
* Absolute neutrophil count > 1,500/mm^3
* Hemoglobin > 9 g/dL
* Platelet count > 100,000/mm^3
* Potassium normal*
* Total calcium (corrected) normal*
* Magnesium normal*
* Phosphorus normal*
* aspartate transaminase (AST) and alanine transaminase (ALT) < 2.5 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN
* Negative proteinuria by dipstick OR total urinary protein ≤ 500 mg with creatinine clearance ≥ 50 mL/min by 24-hour urine collection
* Creatinine < 1.5 times ULN OR creatinine clearance > 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No acute or chronic liver or renal disease
* left ventricular ejection fraction (LVEF) ≥ 45% by Multi Gated Acquisition Scan (MUGA) or echocardiogram
* No complete left bundle branch block
* No obligate use of a cardiac pacemaker
* No congenital long QT syndrome
* No history of or current ventricular or atrial tachyarrhythmias
* No clinically significant resting bradycardia (i.e., heart rate < 50 beats/minute)
* No right bundle branch block with left anterior hemiblock (bifascicular block)
* No uncontrolled hypertension ≥ grade 2, history of labile hypertension, or history of poor compliance with an antihypertensive regimen
* No concurrent unstable angina pectoris or angina pectoris within the past 3 months
* No congestive heart failure (CHF)
* No history of CHF or arrhythmias requiring concurrent digoxin or verapamil
* No acute myocardial infarction within the past 3 months
* No other impaired cardiac function or clinically significant cardiac disease
* No peripheral neuropathy ≥ grade 2
* No unresolved diarrhea ≥ grade 2
* No uncontrolled diabetes
* No active or uncontrolled infection requiring intravenous antibiotics
* No impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of vatalanib, hydroxyurea, and/or everolimus, including any of the following:

  * Ulcerative disease
  * Uncontrolled nausea, vomiting, or diarrhea
  * Malabsorption syndrome
  * Small bowel resection
* No other concurrent severe and/or uncontrolled medical condition that would preclude study participation or compliance
* No known HIV positivity
* No other primary malignancy that is clinically significant or requires active intervention NOTE: *Supplement allowed

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 2 weeks since prior tumor biopsy (4 weeks since prior surgical resection)
* Prior polifeprosan 20 with carmustine implant (Gliadel® wafer) allowed at discretion of principal investigator
* Prior hydroxyurea allowed
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas and 1 week for metronomic-dosed chemotherapy [e.g., daily etoposide hydrochloride or cyclophosphamide]) and recovered
* More than 4 weeks since prior radiotherapy and recovered
* More than 2 weeks since prior immunotherapy and recovered
* More than 4 weeks since prior investigational drugs and recovered
* No prior platelet-derived growth factor- or vascular endothelial growth factor-directed therapies
* More than 2 weeks since prior hematopoietic colony-stimulating factor (e.g., filgrastim [G-CSF] or sargramostim [Granulocyte-macrophage colony-stimulating factor (GM-CSF)])

  * Prior epoetin alfa allowed
* No concurrent warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-07; Primary Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and dose-limiting toxicity of imatinib mesylate and vatalanib when administered with hydroxyurea | 1 Year

SECONDARY OUTCOMES:
Safety | 1.5 Years
Tolerability | 1 Year
Pharmacokinetic | 1.5 Years
  To characterize the single-dose and repeated-dose pharmacokinetic (PK) profiles of imatinib mesylate (in serum) and PTK787/ZK 22584 combination therapy in this patient population.
Antiangiogenic effects | 1 Year
  pre- and post-treatment, of imatinib mesylate, PTK787/ZK 22584 and hydroxyurea combination therapy, using Dynamic contrast enhanced-magnetic resonance imaging (DCE-MRI) to evaluate changes in the extent of vascular permeability, perfusion and relative tumor blood volume; to explore assessment of tumor cellularity and tumor cell death by changes in diffusion weighted imaging magnetic resonance imaging (DWI-MRI) as quantitated by apparent diffusion coefficient maps (ADC maps).
  To note the anti-tumor activity of this regimen in terms of radiographic response, progression-free survival and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: David A. Reardon, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Reardon DA, Egorin MJ, Desjardins A, Vredenburgh JJ, Beumer JH, Lagattuta TF, Gururangan S, Herndon JE 2nd, Salvado AJ, Friedman HS. Phase I pharmacokinetic study of the vascular endothelial growth factor receptor tyrosine kinase inhibitor vatalanib (PTK787) plus imatinib and hydroxyurea for malignant glioma. Cancer. 2009 May 15;115(10):2188-98. doi: 10.1002/cncr.24213. PMID 19248046